CLINICAL TRIAL: NCT07271446
Title: A Phase I, Open-label Study to Evaluate Safety and Tolerability of PB101 in Combination With Standard Treatment, EGFR-TKI, in EGFR-mutated Advanced Non-small Cell Lung Cancer
Brief Title: An Autologous NK/CIK Cell Product (PB101) in Combination With EGFR-TKI for Treating Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Precision Biotech Taiwan Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB-2018-V12
Record Dates: First submitted 2025-09-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: IIIB/IV non-small cell lung cancer; EGFR-TKI combined autologous NK/NKT Cell cell therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Afatinib; osimertinib

STUDY DESIGN:
Intervention Model Description: This study permit standard of care EGFR-TKIs: Gefitinib (Iressa), Erlotinib (Tarceva), Afatinib (Giotrif), or Osimertinib (Tagrisso) will be conducted in one phase. Phase I will investigate safety of PB101. Subjects will be administered 1x10^9＊cells of PB101 over at least 30 minutes weekly for 4 weeks via intravenous infusions, 6 patients will be evaluated. Briefly, after re-visiting to the hospital in 7±3 days to confirm the safety, the subject will continue to be given 1x10^9 cells of PB101 for the following four consecutive weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): This study is designed as an open-label, single-arm Phase I trial to evaluate the safety and tolerability of combining EGFR-TKI therapy with PB101, an autologous NK/NKT cell product. A single-arm design is appropriate for this early-stage investigation because the enrolled patient population consists of individuals with advanced EGFR-mutated NSCLC who have limited treatment options and for whom EGFR-TKI therapy alone often results in eventual acquired resistance. The primary objective at this stage is to assess the safety of adding PB101 to ongoing standard therapy rather than to compare efficacy outcomes between treatment groups.
  Interventions: Biological: PB101 plus EGFR-TKI including gefitinib, erlotinib, afatinib, or osimertinib

INTERVENTIONS:
Biological: PB101 plus EGFR-TKI including gefitinib, erlotinib, afatinib, or osimertinib — This study will be conducted in one phase. Phase I will investigate safety of PB101. Subjects will be administered 1x10^9＊cells (*allow +/-10% cell number) of PB101 over at least 30 minutes weekly for 4 weeks via intravenous infusions, 6 patients will be evaluated. Briefly, after re-visiting to the hospital in 7±3 days to confirm the safety, the subject will continue to be given 1x10^9 cells of PB101 for the following four consecutive weeks.

SUMMARY:
This study was designed to determine the safety and tolerability of PB101 (autologous NK cell product) in combination with standard of care EGFR-TKI in patients with EGFR-mutated advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This study will evaluate the safety of a novel autologous killer cell-based therapeutic product in patients with cancer. The trial targets patients with advanced EGFR-mutated non-small cell lung cancer (NSCLC) who continue EGFR-TKI therapy while receiving PB101-an autologous immune cell product expanded ex vivo and assessed for safety and potential efficacy. The objective is to evaluate the safety and tolerability of PB101 when administered as an adjunct autologous immune-cell therapy.

Autologous natural killer (NK) cells and natural killer T (NKT) cells possess the ability to recognize, remember, and eliminate cancer cells, as well as modulate the functions of other immune cells. Evidence from clinical applications and trials has shown that ex vivo-expanded autologous NK and NKT cells do not produce significant adverse effects and present no major safety concerns when used in cancer therapy. This study will apply our proprietary ex vivo expansion technology for autologous NK and NKT cells to clinically validate the safety and potential therapeutic activity of PB101 in patients with cancer.

This trial will enroll patients with stage III to IV lung cancer. Using our patented technology, autologous immune cells will be isolated and expanded ex vivo for approximately 15 ± 3 days to produce an NK- and NKT-enriched PB101 cell product for adjunctive clinical use. The safety of PB101 will be investigated in a cohort of six participants. Each participant will receive an intravenous infusion of 1 × 10⁹ autologous PB101 cells per dose, followed by a 2-hour post-infusion observation period before discharge. Participants will return for safety assessment 7 ± 3 days after each infusion and will subsequently receive the same dose weekly for a total of four consecutive weeks.

If any participant experiences a CTCAE v5.0 grade ≥3 adverse event during the study, safety data will be reviewed by the Data Safety Monitoring Board (DSMB), and enrollment or continuation of dose administration will proceed only after DSMB confirmation of safety. The presence or absence of adverse reactions among the six participants will determine the safety profile of the cell product and the maximum tolerated dose (MTD). A Phase II trial will be conducted based on Phase I results, expanding cohorts at a confirmed safe dose level to further evaluate clinical efficacy and therapeutic benefit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 20 years of age or older.
* Subjects with histologically or cytologically confirmed stage IIIB/IV non-small cell lung cancer, not amenable to definitive multi-modality therapy, or recurrent disease after a prior diagnosis of stage I-III disease. All staging is via the American Joint Committee on Cancer (AJCC)/IASLC 7th edition proposed staging criteria.
* EGFR sensitizing mutation must be detected in tumor tissue. Specifically, patients harboring the most common mutations, deletions in exon 19 or the L858R mutation in exon 21 are eligible. Other EGFR sensitizing mutations may be eligible after discussion with the principal investigator.
* Subjects must have measurable or evaluable disease according to RECIST v1.1.
* Patients may have had a prior EGFR-TKI including gefitinib, erlotinib, afatinib, or osimertinib in the metastatic setting, but treatment duration must have been less than three months at the time of enrollment.
* Patients may have had no more than one prior line of chemotherapy or immunotherapy in the metastatic setting. At least 14 days must have elapsed from the last chemo/immunotherapy administration until the start of protocol treatment, and patients must have recovered from the side effects of any of these agents.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Acceptable organ function, as evidenced by the following laboratory data:

  1. . Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x upper limit of normal (ULN). (for patients with known hepatic metastases, AST and/or ALT <5x ULN)
  2. . Total serum bilirubin ≤1.5 x ULN
  3. . Absolute neutrophil count (ANC) ≥1500 cells/mm3
  4. . Platelet count ≥75,000 cells/mm3
  5. . Hgb ≥ 10.0 g/dL
  6. . Serum creatinine levels ≤1.5 * ULN, or calculated (by Cockcroft-Gault formula or other accepted formula) or measure creatinine clearance ≥50 mL/min.

Exclusion Criteria:

* Patients with history of clinically significant interstitial lung disease or radiation pneumonitis.
* Patients with brain metastasis or leptomeningeal disease.
* Patients who have had radiation to the lung fields within four weeks of starting treatment. For all palliative radiation to all other sites, at least 7 days must have elapsed prior to starting to treatment.
* Patients who have had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within two weeks prior to starting study drug or who have not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the study ≥1 week after the procedure.
* Patients with a second, clinically active, cancer. Patients with second cancers which have been treated with curative intent and/or are currently inactive are allowed.
* Known history of human immunodeficiency virus (HIV) seropositivity.
* Participants who are receiving any other investigational agents. Patients previously treated with investigational agents must complete a washout period of at least one week or five half-lives, whichever is longer, before starting treatment.
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroid use, except those on topical or inhaled steroids, or steroids given via local injection.
* Patients with clinically significant, uncontrolled cardiovascular disease, such as: unstable angina or myocardial infarction within 6 months prior to screening, abnormal left ventricular ejection fraction (LVEF <50%), cardiac arrhythmia not controlled with medication, uncontrolled hypertension defined as a SBP ≥ 160mm Hg and/or DBP ≥ 100mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
* Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management.
* Pregnancy and lactating women.
* Active hepatitis B or C without treatment.
* Other situations the investigators think not eligible for participation in the research.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Safety assessment by Adverse events (AEs) | From the beginning of the treatment to 1 year after completing 4 doses treatment
  The incidence of adverse events (AEs) was assessed by CTCAE v5.0 including the frequency and type of local toxic reactions at the injection site, including pain, lumps, erythema, granulomas, sterile cysts, and local toxic reactions judged by the clinician.
Safety assessment by Severe Adverse events (SAEs) | From the beginning of the treatment to 1 year after completing 4 doses treatment
  The incidence of severe adverse events (SAEs) was assessed by CTCAE v5.0 including the frequency and type of systemic toxic reactions, nausea, vomiting, fatigue, fever, headache, allergic reactions, uveitis, immune arthritis, and systemic toxic reactions judged by the clinician.

SECONDARY OUTCOMES:
Efficacy assessment by participants' overall response rate (ORR) | From Day -15 before treatment to 1 year after completing 4 doses cell therapy
  The overall response rate (ORR) indicate that the percentage of patients in a clinical trial whose cancer has either completely disappeared or shown a significant reduction in size after treatment
Efficacy assessment by participants' duration of response (DR) | From Day -15 before treatment to 1 year after completing 4 doses cell therapy
  Secondary endpoints included duration of response (DR). Duration of Response (DoR) is a clinical trial endpoint, often used in oncology, measuring the length of time a patient's tumor continues to respond to treatment, from the onset of the response until disease progression or death.
Efficacy assessment by participants' progression-free survival (PFS) | From Day -15 before treatment to 1 year after completing 4 doses cell therapy
  Participants' progression-free survival (PFS) is the length of time that passes from the start of a clinical trial to either the disease getting worse (progression) or the participant dying.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Der Lee, MD PhD, Study Director — Department of Hematology and Oncology, Taipei Medical University Hospital
Locations (1):
- Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Tri-Service General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Q, Liu XY, Zhang T, Zhang XF, Zhao L, Long F, Liu ZK, Wang EH. The dual-functional capability of cytokine-induced killer cells and application in tumor immunology. Hum Immunol. 2015 May;76(5):385-91. doi: 10.1016/j.humimm.2014.09.021. Epub 2014 Oct 8. PMID 25305457
- [Result] Woan K, Reddy V. Potential therapeutic role of natural killer cells in cancer. Expert Opin Biol Ther. 2007 Jan;7(1):17-29. doi: 10.1517/14712598.7.1.17. PMID 17150016
- [Result] Waterhouse P, Penninger JM, Timms E, Wakeham A, Shahinian A, Lee KP, Thompson CB, Griesser H, Mak TW. Lymphoproliferative disorders with early lethality in mice deficient in Ctla-4. Science. 1995 Nov 10;270(5238):985-8. doi: 10.1126/science.270.5238.985. PMID 7481803
- [Result] Ware KE, Hinz TK, Kleczko E, Singleton KR, Marek LA, Helfrich BA, Cummings CT, Graham DK, Astling D, Tan AC, Heasley LE. A mechanism of resistance to gefitinib mediated by cellular reprogramming and the acquisition of an FGF2-FGFR1 autocrine growth loop. Oncogenesis. 2013 Mar 25;2(3):e39. doi: 10.1038/oncsis.2013.4. PMID 23552882
- [Result] Mollet TW, Garcia CA, Koester G. Skin metastases from lung cancer. Dermatol Online J. 2009 May 15;15(5):1. PMID 19624979
- [Result] Thompson CB, Allison JP. The emerging role of CTLA-4 as an immune attenuator. Immunity. 1997 Oct;7(4):445-50. doi: 10.1016/s1074-7613(00)80366-0. No abstract available. PMID 9354465
- [Result] Small EJ, Fratesi P, Reese DM, Strang G, Laus R, Peshwa MV, Valone FH. Immunotherapy of hormone-refractory prostate cancer with antigen-loaded dendritic cells. J Clin Oncol. 2000 Dec 1;18(23):3894-903. doi: 10.1200/JCO.2000.18.23.3894. PMID 11099318
- [Result] Shi SB, Tang XY, Tian J, Chang CX, Li P, Qi JL. Efficacy of erlotinib plus dendritic cells and cytokine-induced killer cells in maintenance therapy of advanced non-small cell lung cancer. J Immunother. 2014 May;37(4):250-5. doi: 10.1097/CJI.0000000000000015. PMID 24714359
- [Result] Sheng J, Fang W, Liu X, Xing S, Zhan J, Ma Y, Huang Y, Zhou N, Zhao H, Zhang L. Impact of gefitinib in early stage treatment on circulating cytokines and lymphocytes for patients with advanced non-small cell lung cancer. Onco Targets Ther. 2017 Feb 21;10:1101-1110. doi: 10.2147/OTT.S112158. eCollection 2017. PMID 28260924
- [Result] Seino K, Motohashi S, Fujisawa T, Nakayama T, Taniguchi M. Natural killer T cell-mediated antitumor immune responses and their clinical applications. Cancer Sci. 2006 Sep;97(9):807-12. doi: 10.1111/j.1349-7006.2006.00257.x. Epub 2006 Jun 29. PMID 16805854
- [Result] Segal NH, Parsons DW, Peggs KS, Velculescu V, Kinzler KW, Vogelstein B, Allison JP. Epitope landscape in breast and colorectal cancer. Cancer Res. 2008 Feb 1;68(3):889-92. doi: 10.1158/0008-5472.CAN-07-3095. PMID 18245491
- [Result] Perez VL, Van Parijs L, Biuckians A, Zheng XX, Strom TB, Abbas AK. Induction of peripheral T cell tolerance in vivo requires CTLA-4 engagement. Immunity. 1997 Apr;6(4):411-7. doi: 10.1016/s1074-7613(00)80284-8. PMID 9133420
- [Result] Parkhurst MR, Riley JP, Dudley ME, Rosenberg SA. Adoptive transfer of autologous natural killer cells leads to high levels of circulating natural killer cells but does not mediate tumor regression. Clin Cancer Res. 2011 Oct 1;17(19):6287-97. doi: 10.1158/1078-0432.CCR-11-1347. Epub 2011 Aug 15. PMID 21844012
- [Result] Ocean AJ, Vahdat LT. Chemotherapy-induced peripheral neuropathy: pathogenesis and emerging therapies. Support Care Cancer. 2004 Sep;12(9):619-25. doi: 10.1007/s00520-004-0657-7. PMID 15258838
- [Result] Niu Q, Wang W, Li Y, Qin S, Wang Y, Wan G, Guan J, Zhu W. Cord blood-derived cytokine-induced killer cells biotherapy combined with second-line chemotherapy in the treatment of advanced solid malignancies. Int Immunopharmacol. 2011 Apr;11(4):449-56. doi: 10.1016/j.intimp.2010.12.014. Epub 2011 Jan 5. PMID 21215350
- [Result] Morgillo F, Della Corte CM, Fasano M, Ciardiello F. Mechanisms of resistance to EGFR-targeted drugs: lung cancer. ESMO Open. 2016 May 11;1(3):e000060. doi: 10.1136/esmoopen-2016-000060. eCollection 2016. PMID 27843613
- [Result] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273
- [Result] Kirkwood JM, Tarhini AA, Panelli MC, Moschos SJ, Zarour HM, Butterfield LH, Gogas HJ. Next generation of immunotherapy for melanoma. J Clin Oncol. 2008 Jul 10;26(20):3445-55. doi: 10.1200/JCO.2007.14.6423. PMID 18612161
- [Result] Kim H, Kim SH, Kim MJ, Kim SJ, Park SJ, Chung JS, Bae JH, Kang CD. EGFR inhibitors enhanced the susceptibility to NK cell-mediated lysis of lung cancer cells. J Immunother. 2011 May;34(4):372-81. doi: 10.1097/CJI.0b013e31821b724a. PMID 21499124
- [Result] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Result] Jordan CT, Guzman ML, Noble M. Cancer stem cells. N Engl J Med. 2006 Sep 21;355(12):1253-61. doi: 10.1056/NEJMra061808. No abstract available. PMID 16990388
- [Result] Jin S, Deng Y, Hao JW, Li Y, Liu B, Yu Y, Shi FD, Zhou QH. NK cell phenotypic modulation in lung cancer environment. PLoS One. 2014 Oct 9;9(10):e109976. doi: 10.1371/journal.pone.0109976. eCollection 2014. PMID 25299645
- [Result] He S, Yin T, Li D, Gao X, Wan Y, Ma X, Ye T, Guo F, Sun J, Lin Z, Wang Y. Enhanced interaction between natural killer cells and lung cancer cells: involvement in gefitinib-mediated immunoregulation. J Transl Med. 2013 Aug 12;11:186. doi: 10.1186/1479-5876-11-186. PMID 23937717
- [Result] Gutierrez-Gutierrez G, Sereno M, Miralles A, Casado-Saenz E, Gutierrez-Rivas E. Chemotherapy-induced peripheral neuropathy: clinical features, diagnosis, prevention and treatment strategies. Clin Transl Oncol. 2010 Feb;12(2):81-91. doi: 10.1007/S12094-010-0474-z. PMID 20156778
- [Result] Fukuoka M, Wu YL, Thongprasert S, Sunpaweravong P, Leong SS, Sriuranpong V, Chao TY, Nakagawa K, Chu DT, Saijo N, Duffield EL, Rukazenkov Y, Speake G, Jiang H, Armour AA, To KF, Yang JC, Mok TS. Biomarker analyses and final overall survival results from a phase III, randomized, open-label, first-line study of gefitinib versus carboplatin/paclitaxel in clinically selected patients with advanced non-small-cell lung cancer in Asia (IPASS). J Clin Oncol. 2011 Jul 20;29(21):2866-74. doi: 10.1200/JCO.2010.33.4235. Epub 2011 Jun 13. PMID 21670455
- [Result] Chang N, Duan J, Wang L, Dong Z, Liu Z. Patients with advanced non-small cell lung cancer with EGFR mutations in addition to complex mutations treated with osimertinib have a poor clinical outcome: A real-world data analysis. Oncol Lett. 2020 Sep;20(3):2266-2272. doi: 10.3892/ol.2020.11801. Epub 2020 Jul 1. PMID 32782544
- [Result] Bour-Jordan H, Esensten JH, Martinez-Llordella M, Penaranda C, Stumpf M, Bluestone JA. Intrinsic and extrinsic control of peripheral T-cell tolerance by costimulatory molecules of the CD28/ B7 family. Immunol Rev. 2011 May;241(1):180-205. doi: 10.1111/j.1600-065X.2011.01011.x. PMID 21488898
- [Result] Boivin JF. Second cancers and other late side effects of cancer treatment. A review. Cancer. 1990 Feb 1;65(3 Suppl):770-5. doi: 10.1002/1097-0142(19900201)65:3+3.0.co;2-8. PMID 2406000
- [Result] Beijers AJ, Jongen JL, Vreugdenhil G. Chemotherapy-induced neurotoxicity: the value of neuroprotective strategies. Neth J Med. 2012 Jan;70(1):18-25. PMID 22271810
- [Result] Baxevanis CN, Gritzapis AD, Tsitsilonis OE, Katsoulas HL, Papamichail M. HER-2/neu-derived peptide epitopes are also recognized by cytotoxic CD3(+)CD56(+) (natural killer T) lymphocytes. Int J Cancer. 2002 Apr 20;98(6):864-72. doi: 10.1002/ijc.10251. PMID 11948464

DOCUMENTS (2):
  • Study Protocol: Study protocol-En (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT07271446/Prot_000.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT07271446/ICF_001.pdf